CLINICAL TRIAL: NCT04311164
Title: Steno Tech Explore: A Multisite Exploratory Study of People With Type 1 Diabetes on Insulin Pump Therapy
Brief Title: Steno Tech Explore: A Study of Insulin Pump Users With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Signe Schmidt, MD, PhD, Researcher, Steno Diabetes Center Copenhagen
Other Study IDs: Steno Tech Explore
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: continous subcutaneous insulin infusion; clinical outcomes; psychological outcomes; educational aspects; preferences; inequality and inequity
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steno Tech Survey Respondents: A cohort of individuals with type 1 diabetes treated with CSII at either SDCC or NOH participating in the Steno Tech Survey.
  Interventions: Other: Questionnaire-based survey
- General Type 1 Diabetes Population: A cohort consisting of the entire population of people with type 1 diabetes in Denmark not included in the Steno Tech Survey cohort (ca. 25.000 individuals).
  Interventions: Other: No intervention given.

INTERVENTIONS:
Other: Questionnaire-based survey — The online questionnaire-based survey is composed of multiple items including pre-coded (multiple choice) questions, dichotomous (yes/no) questions, rating scales and validated questionnaire scales to measure general and diabetes/insulin pump-specific behavior, psychological concepts and preferences.
  Groups: Steno Tech Survey Respondents
Other: No intervention given. — No intervention was given.
  Groups: General Type 1 Diabetes Population

SUMMARY:
The present study is part of an overarching study being conducted in Denmark at Steno Diabetes Center Copenhagen (SDCC) and Nordsjællands Hospital Hillerød (NOH), Steno Tech, that aims to develop and ultimately, in a randomized controlled trial (RCT), test approaches that can assist people with type 1 diabetes in obtaining optimal outcomes using CSII. Through a large-scale, questionnaire-based online survey enriched with data from national registers, this sub-study contributes to this overarching aim by exploring the importance of individual differences across a wide range of factors, including demographic, socioeconomic, health status, psychosocial and preference structures, for optimal use of CSII in people with type 1 diabetes.

DETAILED DESCRIPTION:
See attached protocol for a detailed description.

ELIGIBILITY:
The Steno Tech Survey Repondents group:

* Adult (18+ years)
* Type 1 diabetes
* Insulin pump user
* Danish-speaking

The General Type 1 Population group:

* Adult (18+ years)
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of two groups/cohorts:
  1. Steno Tech Survey Respondents: A cohort of individuals with type 1 diabetes treated with CSII at either Steno Diabetes Center Copenhagen or Nordsjaellands Hospital Hilleroed participating in the Steno Tech Survey.
  2. General Type 1 Diabetes Population: A cohort consisting of the entire population of people with type 1 diabetes in Denmark not included in the Steno Tech Survey cohort (ca. 25.000 individuals).
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin A1c (HbA1c) | 13 years (from 2008 (beginning of register) to present)
  Information on HbA1c in mmol/mol will be extracted from national registers

SECONDARY OUTCOMES:
Other diabetes-relevant biomarkers | 13 years (from 2008 (beginning of register) to present)
  Biomarkers included at the regular diabetes 'check-up' other than HbA1c including hemoglobin, eGFR, UACR, cholesterol total, HDL, LDL, VLDL, triglycerides and TSH will be extracted from national registers
General diabetes and insulin pump-specific behavior | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with single items in the survey
Psychological well-being | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with the WHO5 questionnaire scale in the survey
Diabetes distress | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with the Type 1 Diabetes Distress (T1-DDS) questionnaire scale in the survey
Hypoglycemia anxiety | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with the Hypoglycemia Fear Survey short-form (HFS-SF) questionnaire scale in the survey
Technology-specific satisfaction | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with the Insulin Device Satisfaction Survey (IDSS) and the Glucose Monitoring Satisfaction Survey (GMSS) questionnaire scales in the survey
Educational, time and risk preferences | 1 day (measured at one time point only, i.e., at the survey completion date for each participant)
  Measured with single items in the survey and experimental tasks

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Nordsjællands Hospital Hillerød, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lorenzen JT, Madsen KP, Cleal B, Joensen LE, Norgaard K, Pedersen-Bjergaard U, Schmidt S, Rytter K, Willaing I. Associations between use of diabetes technology and diabetes distress: a Danish cross-sectional survey of adults with type 1 diabetes. BMJ Open. 2024 Mar 25;14(3):e080053. doi: 10.1136/bmjopen-2023-080053. PMID 38531585
- [Derived] Rytter K, Madsen KP, Andersen HU, Hommel E, Pedersen-Bjergaard U, Schmidt S, Norgaard K. Associations between insulin pump self-management and HbA1c in type 1 diabetes. Diabet Med. 2023 Jun;40(6):e15068. doi: 10.1111/dme.15068. Epub 2023 Feb 25. PMID 36786049

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT04311164/Prot_SAP_000.pdf